CLINICAL TRIAL: NCT07010562
Title: A Multi-site, Pre-clinical, Prospective Data Collection Study in Patients Undergoing a Right Heart Catheterization
Status: Not yet recruiting | Type: Observational
Sponsor: Acorai AB (Industry)
Responsible Party: Sponsor
Other Study IDs: Pre-clinical_RHC
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RHC: Patients enrolled for a right heart catheterization procedure as part of their standard of care.
  Interventions: Device: Data collection

INTERVENTIONS:
Device: Data collection — A supervised session that includes 10 minutes of patient information entry, 5 minutes of sensor recording time and 10 minutes of margin for setting up the system and patient, thus a total evaluation duration of approximately 25 minutes prior to the Right Heart Catheterization. No follow-up period for the subjects will be required for this clinical investigation. Patients will be followed as per standard of care, at the hospital. A single follow-up observational data collection will be conducted at 90 days, to collect the number of unplanned hospitalizations since the procedure visit. This does not involve active patient participation.

SUMMARY:
Acorai is developing a non-invasive monitoring system for the estimation of intracardiac hemodynamic parameters in patients with suspected or confirmed heart failure, and/or pulmonary hypertension, who require hemodynamic assessment. The device will be intended as a companion test or clinical decision support tool to be used and interpreted by qualified healthcare professionals to aid standard-of-care clinical assessment in identifying hemodynamic congestion and supporting personalized treatment of heart failure and pulmonary congestion.

This study is part of the development of a non-invasive monitoring system for the estimation of intracardiac hemodynamic parameters. It will be conducted to collect the data needed to train the machine learning models retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age at the time of screening.
* Subject is willing and physically able to comply with the specified evaluations as per the protocol.
* Subject is referred for invasive hemodynamic assessment with right heart catheterization.
* Subject has provided written informed consent using the approved consent form.

Exclusion Criteria:

* Discretionary exclusion when the inclusion of a potential subject is not in their best interest or not in the interest of compliant performance of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled for a right heart catheterization procedure as part of their standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 392 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the ML's performance to estimate pressure | Day 0 to Day 90
  Performance of the Machine Learning model trained on data collected from the device to estimate left-sided filling pressure compared to right heart catheterization.